CLINICAL TRIAL: NCT01007812
Title: Clinical Comparison of Two Silicone Hydrogel Toric Lenses in the US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P-242-C-032
Record Dates: First submitted 2009-11-02; First posted 2009-11-04 (Estimated); Results first posted 2010-11-17 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-01

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Lotrafilcon B / Comfilcon A (Other): Lotrafilcon B silicone hydrogel, toric, soft contact lenses worn for one week, followed by Comfilcon A silicone hydrogel, toric, soft contact lenses worn for one week.
  Interventions: Device: Lotrafilcon B contact lens; Device: Comfilcon A contact lens
- Comfilcon A / Lotrafilcon B (Other): Comfilcon A silicone hydrogel, toric, soft contact lenses worn for one week, followed by Lotrafilcon B silicone hydrogel, toric, soft contact lenses worn for one week.
  Interventions: Device: Lotrafilcon B contact lens; Device: Comfilcon A contact lens

INTERVENTIONS:
Device: Lotrafilcon B contact lens — Silicone hydrogel, toric, soft contact lens
Device: Comfilcon A contact lens — Silicone hydrogel, toric, soft contact lens

SUMMARY:
The purpose of this trial is to compare the performance of two different contact lenses for contact lens wearers with astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Have a current spectacle prescription, preferably within 6-9 months.
* Currently wearing toric soft contact lenses in both eyes with at least 1 month experience wearing current brand for daily wear.
* Be correctable to at least 20/40 distance visual acuity in each eye while wearing trial lenses in the parameters available for this trial.
* Have acceptable or optimal fit for each eye at the dispense of each pair of study lenses.
* Other protocol-defined inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks immediately prior to enrollment for this trial.
* Currently enrolled in any Clinical Trial.
* Evidence of systemic or ocular abnormality, infection or disease which is likely to affect successful wear of contact lenses or use of their accessory solutions as determined by the investigator.
* Any use of medications for which contact lens wear could be contraindicated as determined by the investigator.
* Currently wearing soft toric contact lenses as extended wear.
* Currently wearing either of the products to be worn in the study.
* Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Lotrafilcon B / Comfilcon A: Lotrafilcon B silicone hydrogel, toric, soft contact lenses worn for one week, followed by Comfilcon A silicone hydrogel, toric, soft contact lenses worn for one week. Both products worn in a daily wear modality.
- Comfilcon A / Lotrafilcon B: Comfilcon A silicone hydrogel, toric, soft contact lenses worn for one week, followed by Lotrafilcon B silicone hydrogel, toric, soft contact lenses worn for one week. Both products worn in a daily wear modality.
Period: Period 1, One Week
Arm/Group | Lotrafilcon B / Comfilcon A | Comfilcon A / Lotrafilcon B
Started | 25 | 25
Completed | 24 | 24
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Discomfort | 1 | 0
Period: Period 2, One Week
Arm/Group | Lotrafilcon B / Comfilcon A | Comfilcon A / Lotrafilcon B
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: This reporting group includes all enrolled and dispensed subjects.
Arm/Group | Overall Study
Number analyzed (Participants) | 50
Age Continuous [Mean (Standard Deviation); unit: years] | 33.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Vision
Description: Overall vision, as interpreted by the subject and reported by the subject on a questionnaire as a single, retrospective evaluation of one week's wear time. Overall vision was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: After 1 week of wear
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B Contact Lens | Comfilcon A Contact Lens
Number analyzed (Participants) | 48 | 48
Units on a Scale | 8.2 (1.8) | 8.3 (1.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 29 days.
Description: In this cross-over study, each participant wore the first product per the randomization, but not the second, due to discontinuation from the study.
Arm/Group | Lotrafilcon B Contact Lens | Comfilcon A Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.